CLINICAL TRIAL: NCT02451449
Title: Celiac Disease and Infertility Among Men and Women in Denmark: Prevalence of Celiac Disease Among Men and Women Treated in Danish Public Fertility Clinics
Brief Title: Celiac Disease and Infertility Among Men and Women in Denmark
Acronym: CØF2015
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: CØF 2015
Record Dates: First submitted 2015-02-17; First posted 2015-05-22 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2017-10

CONDITIONS: Celiac Disease; Infertility
Keywords: Celiac disease; Infertility; Prevalence study
MeSH Terms: conditions — Celiac Disease; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood Biopsy of small-bowel
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to estimate the prevalence of celiac disease in a population of men and women newly referred to fertility treatment in Danish public fertility clinics.

DETAILED DESCRIPTION:
Aims of the study:

* To investigate the prevalence of CD in a cohort of men and women referred to fertility treatment in Danish fertility clinics
* To compare individuals diagnosed with CD to individuals without the disease to investigate:

  * possible predictive symptoms of CD (fertility history, gastrointestinal symptoms, co-morbidity)
  * semen quality among men
* To investigate the effect of a gluten free diet on semen quality (DNA fragmentation) in men diagnosed with CD before and after 3 months treatment with a gluten free diet
* To investigate correlation between sCD163 and histological changes in the small-bowel
* To investigate the correlation between level of sCD163 and level of macrophages in biopsies
* To evaluate the performance of a rapid point-of-care serologic CD screening test in a population of men and women referred to fertility treatment

Hypothesises of the study:

* CD increases the risk of infertility in both men and women
* Predictive symptoms of CD can be identified and used to select future risk-groups
* Untreated CD in men has a negative effect on semen quality and semen quality improves by treatment with a gluten free diet
* Level of sCD 163 correlates with degree of inflammatory lesions in the small-bowel
* Level of sCD163 correlate with level of macrophages in the mucose-tissue of the small-bowel
* The rapid point-of-care test is an efficient tool for CD case finding in an adult population

Methods and materials:

A cross-sectional study measuring the prevalence of Celiac disease in a population of couples (men and women) referred to treatment in Danish fertility clinics. Analysis of data from study questionnaires, serological tests, semen specimens and small-bowel biopsies will be performed and one year follow-up on fertility treatment outcome of all participants.

Recruitment:

A realistic sample size to recruit in 2 years is 600 women and 600 men (600 heterosexual couples) newly referred to two Danish public fertility clinics. Both the male and female part will be asked to participate when they attend the clinic for pre-assessment. Patients with a prior biopsy confirmed CD will not be screened, but will count in the prevalence result.

Questionnaires:

After giving informed consent patients will be asked to answer a questionnaire about gastrointestinal function (The Gastrointestinal Symptom Rating Scale, GSRS (26)), fertility history and co-morbidity (appendix I). The GSRS questionnaire is a validated, self-administered questionnaire that includes 15 questions, which assess severity of gastrointestinal symptoms using a 7-point Likert scale in five domains: indigestion, diarrhoea, constipation, abdominal pain and reflux. The severity of symptoms reported in the GSRS increases with increasing score.

Serological tests:

After answering the questionnaire a blood sample will be drawn and send to the laboratory and analysed for IgA Antitissue Transglutaminase (IgA TG ), total IgA and IgG Deamidated Gliadin Peptid (DGP) if IgA deficit and sCD163. At the same time an in vitro rapid screening test for CD will be performed (Simtomax®). Simtomax® will indicate CD and IgA deficiency (based on Deamidated Gliadin Peptid and total IgA). The cut off value for CD positive tests and referral to gastroscopy with small- bowl biopsy is IgA TG > 7 kU/L and for the Simtomax® the test results "celiac positive IgA normal" and "celiac positive IgA deficient" together with clinical symptoms (questionnaire). For Total IgA cut off value is < 0,80 g/L. Simtomax® has a high negative predict value (>90%) on CD. The cut off value for IgG DGP is > 3 KU/L. One CD positive test is enough for referral to small-bowel biopsy.

Level of sCD163 will be measured but level of sCD163 has no consequence for further referral or diagnose of CD.

All serological tests will be sent to Department of Biochemistry at Horsens Hospital, who is responsible of handling all serological tests in this study. Serological material will be destroyed immediately after analysis.

Follow-up algorithm after serological tests:

* Patients, who tests negative for CD in IgA TG, IgG DGP and Simtomax® will, by telephone or consultation in the fertility clinic, be informed by the study nurse or doctor of the results. Results will be available within 5 days. The patients will continue fertility treatment as planned.
* If IgA TG or IgG DGP (or Simtomax® with clinical symptoms) exceeds the cut off value, indicating CD, the patient will be contacted by the investigator and informed of the results and invited to a consultation and gastroscopy by the responsible specialist doctor at Department of Endoscopy, Horsens Hospital. The patient will receive verbal and written information about preparation before gastroscopy and risk and complications of the procedure and small-bowel biopsy.

The biopsy material will be send to pathology analysis to determine histology classification (Marsh-classification).

Small-bowel biopsy:

Biopsies will be taken from the small-bowel (duodenum and duodenal bulb 5-6 biopsies). The classic pathology changes of CD in the small-bowel are categorised by the "Modified Marsh criteria" determining the histological changes:

* Marsh stage 0: normal duodenal mucosa
* Marsh stage 1: increased number of intra-epithelial lymphocytes (IELs), usually exceeding 25 per 100 enterocytes
* Marsh stage 2: Stage 1 + crypt hyperplasia
* Marsh stage 3 (a,b,c): Increased IELs, crypt hyperplasia and partial, subtotal or total villous atrophy A Marsh stage 3 (a,b,c) is the classic lesions of CD and confirms a diagnose of CD. Stage 1 and 2 is indicating milder lesions of the small-bowel, indicating CD. A Marsh 0 but positive serology are rare but may indicate latent CD. Patients with a Marsh 0 classified biopsy will not be classified as having CD. Patients with 1-3 (a,b,c) classified biopsy and elevated IgA TG or IgG DGP will in this study be considered as having CD (27).

Levels of sCD163 will be compared with Marsh stage to determine if levels of sCD 163 correlate with the inflammatory lesion of the small-bowel.

Biopsies will, after determination of Marsh stage, undergo coloring to identify macrophages. Biopsies will be destroyed at study end.

Follow-up algorithm after biopsy:

The patient will be informed of the pathology answer by telephone by the responsible specialist doctor and be offered follow-up according to this algorithm:

* Patients with positive serology but negative biopsy will be offered a consultation with a specialist doctor at Horsens Hospital.
* Patients with biopsy confirmed CD will be offered consultation with a specialist doctor and dietary counselling by a hospital dietician at Horsens Hospital
* Patients with a biopsy confirmed CD will be offered new consultation in the fertility clinic planning their further fertility treatment (they are recommended a strict gluten free diet of at least three months before fertility treatment take place (both male and female patients).
* Patients with a biopsy confirmed CD will be offered three month follow-up with a specialist doctor at Horsens Hospital. Here the patient will be asked to answer the second part of the questionnaire again, new serological tests (IgA TG, IgG DGP, sCD163) and male patients to deliver a new semen specimen.

Semen specimens:

All male patients will as a routine procedure deliver semen specimens for semen quality analysis (based on motility, morphology, semen concentration) at consultation in the fertility clinics. This study uses the results from the routine semen quality analysis for all male participants.

Men with a biopsy confirmed CD will be asked to collect a semen specimen before starting on a gluten free diet and to collect a semen specimen again after 3 months on a gluten free diet. These semen specimens will be frozen and tested for chromatin fragmentation. The semen quality is measured by the degree of chromatin fragmentation within the sperm cell using Sperm Chromatin Structure Assay (SCSA). Semen quality is expressed in a DNA fragmentation index, expressing the percent of damaged sperm. The before and after gluten free diet DNA fragmentation index will be compared.

Biobank for future research:

This study contains a biobank. Patients will be asked to give separate informed consent to store blood material in a biobank for future research. If they consent, one extra glass of 10 ml full blood will be drawn at inclusion, and for patients diagnosed with CD also one extra glass of 10 ml at 3 months follow-up. The Danish Data Protection Agency has given permission to establish a biobank. The biobank is for future research and material can only be used with new permission from a regional committee on health research ethics.

Statistics and power calculation:

All data will be analysed using STATA 13.To calculate sample size the formula n= Z2P(1-P)/d2 (24) is used: With a confidence interval (CI) of 95% (Z=1.96), precision of 1% (d=0.01) and an expected prevalence for women of 2,5% (P=0.025), the minimum sample size required is 600 women. For men with P=0.01 and d=0.005 sample size =1521 with CI of 95%. With expected prevalence for couples: (1-(0.975*0.99)) = 3.5% and d=0.0175, CI 95%, sample size = 420 couples.

Ethical considerations:

Participants included in this study could benefit directly from the study if they have an undiagnosed CD. It is evident that an untreated CD in women can have negative consequences in pregnancy. The risk of drawing blood is minimal. If blood tests are indicating CD the risk of actually having CD is more than 50%. Undergoing small-bowel biopsy is unpleasant but not painful. It is a standard procedure. Participants will be informed of risks before consenting. Clinical advisor, senior consultant in gastroenterology Thomas Møller Jensen, Horsens Hospital is responsible for the medical and clinical management and follow-up of patients detected with CD positive serological test. The approval from the Regional Committee on Health Research Ethics, Central Denmark and The Danish Data Protection Agency has been obtained before study start. The study will be carried out in accordance with the Helsinki II declaration and oral and written informed consent will be obtained from all patients participating. Consent to store blood in a biobank for future research is given separately. The processing of data is in accordance with the Danish regulation. All information will be kept confidentially and locked up in the fertility clinics until data are collected by investigator and then kept locked up (double lock) in the Department at Horsens Hospital. At the end of the study all identifiable personal data will be concealed in a code only accessible by investigator who is also responsible of the biobank.

Funding:

Department of Medicine, Horsens Hospital has taken initiative to this study. There is no economical incentive related to this study for any of the project participants.

The Simtomax® in vitro test will be funded by the pharmaceutical company Tillotts Pharma (1200 tests). The agreement has been authorized through The Technology Transfer Office at Aarhus University. A deficit guarantee on salary to investigator Louise Grode has been given by Horsens Hospital before study start. All costs will be sought funded by private and public funding. A research account administered by Horsens Hospital will hold any funding related to the study.

No payment is given to patients participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women referred to fertility treatment in a fertility clinic in Denmark, (couples)
* Age > 18 years
* Able to read and understand the Danish language

Exclusion Criteria:

* Lack of capacity to consent for themselves
* Individuals not living in Denmark
* Single women
* Homosexual couples

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Both female and male participants are being studied
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2015-01; Primary Completion 2017-09 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of celiac disease | Referral to fertility clinics over a period of two years
  Celiac disease confirmed by histological lesions of the small-bowel

SECONDARY OUTCOMES:
Gastrointestinal symptoms of undiagnosed celiac disease | One week symptoms
  Questionnaire on gastrointestinal symptoms
Soluble CD163 mg/L | baseline
  Inflammatory marker in macrophage activation

OTHER OUTCOMES:
Semen quality in celiac disease | baseline and after 3 months glutenfree treatment
  Chromatin structure

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Ramlau-Hansen, PhD, Study Chair — University of Aarhus
Locations (2):
- Denmark (2):
  - Fertility Clinic, Horsens Hospital, Horsens, Central Jutland
  - Fertility Clinic, Skive Hospital, Skive, Central Jutland

IPD SHARING:
Plan to Share IPD: No